CLINICAL TRIAL: NCT03520907
Title: The Effect of the Transversalis Fascia Plane Block on Postoperative Pain Behavior After Hernia Repair Surgery in Children - Comparison With Conventional Ilioinguinal/Iliohypogastric Nerve Block-
Brief Title: The Comparison of the Transversalis Fascia Plane Block With Ilioinguinal/Iliohypogastric Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kazuhiko Okuyama, MD (Other)
Responsible Party: Sponsor-Investigator, Kazuhiko Okuyama, MD, Chief Anesthesiologist, Ibaraki Children's Hospital
Organization: Ibaraki Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TFPBvsIIB
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Pain; Inguinal Hernia Unilateral; Children, Only
Keywords: transversalis fascia; ilioinguinal/iliohypogastric nerve; inguinal hernia repair; children
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascia Plane Block (Experimental): receive transversalis fascia plane block with 0.4 ml/kg of 0.25% levobupivacaine after establishment of general anesthesia.
  Interventions: Drug: Transversalis Fascia Plane Block
- Ilioinguinal/iliohypogastric Nerve Block (Active Comparator): receive ilioinguinal/iliohypogastric nerve block with 0.1 ml/kg of 0.25% levobupivacaine after establishment of general anesthesia.
  Interventions: Drug: Ilioinguinal/iliohypogastric Nerve Block

INTERVENTIONS:
Drug: Transversalis Fascia Plane Block — block will be performed under real-time ultrasound guidance
  Other Names: TFPB
  Arms: Transversalis Fascia Plane Block
Drug: Ilioinguinal/iliohypogastric Nerve Block — block will be performed under real-time ultrasound guidance
  Other Names: II/IH B
  Arms: Ilioinguinal/iliohypogastric Nerve Block

SUMMARY:
This study compares the transversalis fascia plane block with the ilioinguinal/iliohypogastric nerve block in children undergoing hernia repair surgery.

Half of participants will receive the transversalis fascia plane block, while the other will receive the ilioinguinal/iliohypogastric nerve block.

DETAILED DESCRIPTION:
The ilioinguinal/iliohypogastric nerve block (II/IH B)is a widely used regional anesthesia technique in inguinal hernia repair surgery. However, this block provides limited analgesia during and after surgery, and the patients feel pain when walking. The transversalis fascia plane block (TFPB) is a recently developed technique and several case reports presented its efficacy for inguinal repair surgery in adult patients. It may block not only ilioinguinal and iliohypogastric nerves but also splanchnic nerves, which is conveyed via the thoracolumbar fascia. Therefore, we compare the effect of the TFPB and II/IH B on postoperative pain and walking form.

ELIGIBILITY:
Inclusion Criteria:

* the patients undergoing unilateral open hernia repair surgery

Exclusion Criteria:

* known allergy to local anesthetics, psychomotor retardation, anti-epileptic drugs usage, anti-inflammatory drug usage

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
walking appearance | 3 to 5 hours after surgery
  scoring a way of walking; 0: brisk walk, big step, able to skip (= no pain) to 5: not able to stand up ( = worst pain)

SECONDARY OUTCOMES:
FLACC (face, legs, activity, cry, consolability) score | 3 to 5 hours after surgery
  behavioral pain scale in children. Each category has 0 to 2 score; Total 0 (no pain) to 10 (worst)
Faces Pain Scale revised | 3 to 5 hours after surgery
  self-reported pain score. Children choose a face from six faces.
additional pain curer usage | up to 5 hours after surgery
  request or necessity of administration of acetaminophen or flurbiprofen

OTHER OUTCOMES:
intraoperative heart rate changes | just before surgery start, one minute after incision, maximum value during surgery
  heart rate during surgery
intraoperative respiratory rate changes | just before surgery start, one minute after incision, maximum value during surgery
  respiratory rate during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiko Okuyama, MD, Study Director — Ibaraki Children's Hospital
Locations (1):
- Ibaraki Children's Hospital, Mito, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No